CLINICAL TRIAL: NCT03331796
Title: Noninvasive Cortical Stimulation to Improve Memory in Mild Cognitive Impairment
Brief Title: Noninvasive Brain Stimulation for Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Joy Taylor, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAY0003AGG; R01AG055526 (NIH)
Record Dates: First submitted 2017-09-18; First posted 2017-11-06 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment; Mild Neurocognitive Disorder; Cognitive Decline; Mental Deterioration; Cognitive Dysfunction; Memory Decline; Memory Loss; Memory Impairment
Keywords: mild cognitive impairment; tms; rtms; transcranial magnetic stimulation; noninvasive brain stimulation; non-pharmacological
MeSH Terms: conditions — Cognitive Dysfunction; Neurocognitive Disorders; Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Active repetitive transcranial magnetic stimulation (rTMS) (Bilateral DLPFC) (Experimental): One-third of participants will receive active rTMS to the right and left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Active rTMS (Bilateral DLPFC)
- Active repetitive transcranial magnetic stimulation (rTMS) (Bilateral LPC) (Experimental): One-third of participants will receive active rTMS to the right and left lateral parietal cortex (LPC).
  Interventions: Device: Active rTMS (Bilateral LPC)
- Placebo repetitive transcranial magnetic stimulation (rTMS) (Inactive) (Placebo Comparator): One-third of participants will receive placebo/inactive rTMS, either to the DLPFC or the LPC. Those receiving placebo rTMS will serve as the control group.
  Interventions: Device: Placebo rTMS (Inactive)

INTERVENTIONS:
Device: Active rTMS (Bilateral DLPFC) — TMS Stimulation Parameters for the active DLPFC rTMS intervention group will be: 10 Hz, 4-second train duration and 11-second inter-train interval. During each session, 2,000 pulses will be applied for each hemisphere (for a total of 4,000 pulses per session). Participants will receive 20 sessions (1 or 2 sessions per day, M-F).
  Arms: Active repetitive transcranial magnetic stimulation (rTMS) (Bilateral DLPFC)
Device: Active rTMS (Bilateral LPC) — TMS Stimulation Parameters for the active LPC rTMS intervention group will be: 10 Hz, 4-second train duration and 11-second inter-train interval. During each session, 2,000 pulses will be applied for each hemisphere (for a total of 4,000 pulses per session). Participants will receive 20 sessions (1 or 2 sessions per day, M-F).
  Arms: Active repetitive transcranial magnetic stimulation (rTMS) (Bilateral LPC)
Device: Placebo rTMS (Inactive) — For the Placebo rTMS (Inactive) group, the participant will wear scalp electrodes through which a low voltage, low electric current (2-20mA at no more than 100V) is passed to mimic the sensation of receiving actual rTMS. Participants will receive 20 sessions (1 or 2 sessions per day, M-F).
  Arms: Placebo repetitive transcranial magnetic stimulation (rTMS) (Inactive)

SUMMARY:
The goal of this study is to test the efficacy of repetitive Transcranial Magnetic Stimulation (rTMS) as a treatment for Mild Cognitive Impairment (MCI). Participants will be randomly assigned to one of three treatment groups: Group 1: Active Dorsolateral Prefrontal Cortex (DLPFC) rTMS; Group 2: Active Lateral Parietal Cortex (LPC) rTMS; and Group 3: Inactive rTMS (Placebo) control (evenly split between each coil location). Participation in the study takes approximately 7 ½ months-including a 2-to 4-week treatment phase (20 rTMS sessions) and a 6-month follow-up phase.

DETAILED DESCRIPTION:
This study aims to test the efficacy of a non-pharmacological treatment for MCI that involves noninvasive brain stimulation (NIBS). Early studies in Alzheimer's disease (AD) dementia patients have found that repetitive transcranial magnetic stimulation (rTMS, a form of NIBS) improved global cognitive function and activities of daily living. Given that in AD, neuronal loss and synaptic dysfunction progress along brain networks, the results of these early studies of brain stimulation suggest there is sufficient neuroplasticity in AD for efficacious effects of brain stimulation. Of the very few rTMS studies in MCI that have been published, the effect size appears to be moderately large. However, it is not clear whether the dorsolateral prefrontal cortex (DLPFC), the stimulation site used in the most of the prior MCI/AD rTMS trials, is the optimal site for achieving the most efficacious effects including effects on episodic memory. Importantly, when other investigators used rTMS to stimulate a lateral parietal cortical (LPC) site in healthy young adults, significant effects of rTMS on memory were measureable weeks later. Moreover, functional connectivity of brain regions was selectively increased, including the posterior cingulate cortex (PCC), a "hub" of brain networks that is affected in amnestic MCI.

Because stimulation of the DLPFC and the LPC may each have distinct effects, we designed this pilot trial to have two active rTMS treatment groups: DLPFC and LPC. A third group will receive inactive (placebo) rTMS to achieve a controlled, randomized, double-blind trial. For each of the three groups, stimulation will be bilateral, based on effects achieved in the AD studies. The primary hypothesis is that active rTMS (to either site of stimulation) will be superior to inactive (placebo) rTMS in improving memory. Measures of change in functional connectivity will be computed to examine whether there is evidence that rTMS changes connectivity of the PCC with other regions of the brain. In addition to looking at effects of rTMS on functional connectivity and cognition in relation to the cortical site stimulated, genetic markers will be collected toward addressing heterogeneity of response. To track the durability of rTMS effects on memory, participants will be followed longer than in any prior study (up to 6 months after the intervention). If this study finds rTMS improves memory in older adults with MCI, further clinical development of this non-pharmacological treatment could ultimately improve the lives of millions of older adults who have MCI and are at an increased risk of developing dementia.

ELIGIBILITY:
* Both Veterans and Non-Veterans may enroll if they meet the following criteria **

Inclusion Criteria:

* Diagnosed with amnestic Mild Cognitive Impairment (aMCI);
* Stable medications (including any dementia-related meds) for at least 4 weeks prior to Baseline;
* Geriatric Depression Scale score less than 6;
* Ability to obtain a motor threshold, determined during the screening process;
* Study partner available; living situation enables attendance at clinic visits;
* Visual and auditory acuity adequate for neuropsychological testing;
* Good general health with no diseases expected to interfere with the study;
* Participant is not pregnant or of childbearing potential (i.e. women must be 2 years post-menopausal or surgically sterile);
* Modified Hachinski Ischemic score less than or equal to 4;
* Agree to DNA extraction for single nucleotide polymorphism (SNP) genotyping;
* Able to understand study procedures and comply with them for the entire length of the study.

Exclusion Criteria:

* Prior exposure to rTMS within the past 12 months;
* Magnetic field safety concern such as a cardiac pacemaker, cochlear implant, implanted device in the brain (deep brain stimulation), or metal fragments or foreign objects in the eyes, skin or body;
* Any significant neurological disease other than suspected incipient Alzheimer's disease;
* Unstable cardiac disease or recent (< 3 months previous) myocardial infarction. Any significant systemic illness or unstable medical condition that could lead to difficulty with protocol adherence;
* History of epilepsy or repetitive seizures, as determined by patient report or chart review;
* History of a medical condition or current use/abuse of medications and substances that increase the risk of a seizure, specifically:

  * Traumatic brain injury within 2 months that would increase the risk for seizure;
  * Unable to safely withdraw, at least 4 weeks prior to Baseline, from medications that substantially increase the risk of having seizures (for example: theophylline, clozapine, and methylphenidate).
  * Current or past history of a mass lesion, cerebral infarct, or other noncognitive active neurological disease that would increase the risk for seizure.
  * Stimulant abuse within the previous 90 days. Cocaine and abuse of amphetamine and methylphenidate are associated with an increased risk of seizures;
* Major depression or bipolar disorder (DSM-IV) within the past 1 year, or psychotic features within the last 3 months that could lead to difficulty with protocol adherence;
* Taking sedative hypnotics or medications with anti-cholinergic properties and unable to withdraw at least 4 weeks prior to Baseline;
* Current alcohol or substance abuse (not including caffeine or nicotine) within the past 1 year, as determined by chart review, participant or study partner report, or greater than "moderate" alcohol use defined by the Quantity-Frequency-Variability Index (Cahalan, Cisin, & Crossley, 1969);
* Any contraindications for magnetic resonance imaging (MRI) studies, e.g. severe claustrophobia, weight above 350 lb maximum allowed by MRI scanner, pregnancy;
* Participation in another concurrent clinical trial;
* Inability or unwillingness of individual or legal representative to give written informed consent.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy L Taylor, Ph.D., Principal Investigator — Stanford/VA Aging Clinical Center
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liao X, Li G, Wang A, Liu T, Feng S, Guo Z, Tang Q, Jin Y, Xing G, McClure MA, Chen H, He B, Liu H, Mu Q. Repetitive Transcranial Magnetic Stimulation as an Alternative Therapy for Cognitive Impairment in Alzheimer's Disease: A Meta-Analysis. J Alzheimers Dis. 2015;48(2):463-72. doi: 10.3233/JAD-150346. PMID 26402010
- [Derived] Taylor JL, Hambro BC, Strossman ND, Bhatt P, Hernandez B, Ashford JW, Cheng JJ, Iv M, Adamson MM, Lazzeroni LC, McNerney MW. The effects of repetitive transcranial magnetic stimulation in older adults with mild cognitive impairment: a protocol for a randomized, controlled three-arm trial. BMC Neurol. 2019 Dec 16;19(1):326. doi: 10.1186/s12883-019-1552-7. PMID 31842821

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the Stanford/VA Aging Clinical Research Center over a 4-year period, which included a 13-month hiatus during the Coronavirus disease (COVID-19) pandemic. The study was open for recruitment on 05/16/2018. The first participant was enrolled and randomized on 06/15/2018; the last participant was enrolled and randomized on 11/22/2022.
Pre-assignment Details: Of 69 consented, screened participants, 40 participants met inclusion/exclusion criteria and were randomized to treatment.
  This was a dyad study, such that each amnestic Mild Cognitive Impairment (aMCI) participant who enrolled in the study had a study partner whose role was to provide collateral data about the primary participant's everyday functioning. Study partners were not assessed for outcomes such as caregiver burden; therefore, the study partners are not considered enrolled.
Groups:
- Active rTMS (Bilateral DLPFC): One-third of participants will receive active repetitive transcranial magnetic stimulation (rTMS) to the right and left dorsolateral prefrontal cortex (DLPFC).
  Active rTMS (Bilateral DLPFC): Stimulation Parameters for the active DLPFC rTMS intervention group will be: 10 Hz, 4-second train duration and 11-second inter-train interval. During each session, 2,000 pulses will be applied for each hemisphere (for a total of 4,000 pulses per session). Participants will receive 20 sessions (1 or 2 sessions per day, M-F).
- Active rTMS (Bilateral LPC): One-third of participants will receive active rTMS to the right and left lateral parietal cortex (LPC).
  Active rTMS (Bilateral LPC): Stimulation Parameters for the active LPC rTMS intervention group will be: 10 Hz, 4-second train duration and 11-second inter-train interval. During each session, 2,000 pulses will be applied for each hemisphere (for a total of 4,000 pulses per session). Participants will receive 20 sessions (1 or 2 sessions per day, M-F).
- Placebo rTMS (Inactive): One-third of participants will receive placebo/inactive rTMS, either to the DLPFC or the LPC. Those receiving placebo rTMS will serve as the control group.
  Placebo rTMS (Inactive): For the Placebo rTMS (Inactive) group, the participant will wear scalp electrodes through which a low voltage, low electric current (2-20mA at no more than 100V) is passed to mimic the sensation of receiving actual rTMS. Participants will receive 20 sessions (1 or 2 sessions per day, M-F).
Period: Allocation and Primary Endpoint
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Started (40 dyads started the study.) | 14 | 13 | 13
Completed (Of the 40 dyads that started the study, 33 dyads completed Period 1. Not completing Period 1 were 3 dyads and an additional 4 study partners who declined to provide further data about the primary participant. In all, 37 Primary Participants and 33 Study Partners competed Period 1.) | 14 | 12 | 11
Not Completed | 0 | 1 | 2
Not completed — Pandemic Disruption | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Extended Follow-up
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Started (A total of 37 primary participants and 33 Study Partners started Period 2. Of the 37 primary participants, 33 were part of a dyad. The other 4 participants had no one to complete questionnaires about his/her everyday functioning) | 14 | 12 | 11
Completed (Of the 33 dyads that started Period 2, 28 dyads completed. Not completing Period 2 were: 3 dyads; 2 additional study partners who declined to provide further data about the primary participant; and 2 of the 4 participants who entered Period 2 without a study partner. In all, 32 primary participants and 28 Study Partners completed the study.) | 12 | 11 | 9
Not Completed | 2 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Termination of Funding | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The population analyzed included all participants who received at least 1 session of the intervention and who provided primary outcome data post-baseline.
Groups:
- Active rTMS (Bilateral DLPFC): One-third of participants will receive active rTMS to the right and left dorsolateral prefrontal cortex (DLPFC).
  Active rTMS (Bilateral DLPFC): TMS Stimulation Parameters for the active DLPFC rTMS intervention group will be: 10 Hz, 4-second train duration and 11-second inter-train interval. During each session, 2,000 pulses will be applied for each hemisphere (for a total of 4,000 pulses per session). Participants will receive 20 sessions (1 or 2 sessions per day, M-F).
- Active rTMS (Bilateral LPC): One-third of participants will receive active rTMS to the right and left lateral parietal cortex (LPC).
  Active rTMS (Bilateral LPC): TMS Stimulation Parameters for the active LPC rTMS intervention group will be: 10 Hz, 4-second train duration and 11-second inter-train interval. During each session, 2,000 pulses will be applied for each hemisphere (for a total of 4,000 pulses per session). Participants will receive 20 sessions (1 or 2 sessions per day, M-F).
- Total: Total of all reporting groups
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive) | Total
Number analyzed (Participants) | 14 | 12 | 11 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (5.8) | 75.7 (7.5) | 74.0 (5.3) | 74.4 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 16
  Male | 9 | 6 | 6 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 12 | 10 | 11 | 33
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 10 | 8 | 9 | 27
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 11 | 37
Education [Mean (Standard Deviation); unit: years] | 17.0 (2.7) | 16.9 (2.2) | 17.1 (2.5) | 17.0 (2.4)
Mild Cognitive Impairment Stage [Count of Participants; unit: Participants] — Mild Cognitive Impairment Stage (early or late), according to the classification scheme of the Alzheimer's Disease Neuroimaging Initiative (ADNI3)
  Participants
    Early | 6 | 7 | 5 | 18
    Late | 8 | 5 | 6 | 19
Clinical Dementia Rating Scale Sum of Boxes Score [Mean (Standard Deviation); unit: units on a scale] — The Clinical Dementia Rating Scale (CDR)-Sum of Boxes (SOB) score is a continuous measure of dementia severity. Six domains of functioning are covered during interviews with participants and informants: Memory; Orientation; Judgment and problem solving; Community affairs; Home and hobbies; and Personal care. The interviewer rates each domain on a scale that indicates the severity of impairment: 0 = No Impairment, 0.5 = Questionable, 1 = Mild, 2 = Moderate, and 3 = Severe. The CDR-SOB score is the sum of the ratings.
  The CDR-SOB ranges from 0 to18; a higher value reflects a worse outcome.
  units on a scale | 1.3 (0.7) | 1.0 (0.5) | 1.1 (0.6) | 1.1 (0.6)
Logical Memory II subscale (Delayed Recall, Story A only) [Mean (Standard Deviation); unit: units on a scale] — The Logical Memory II - Story A (Anna Thompson) Delayed Recall measure was used to assess verbal memory performance at the Screening visit. The story's text is divided into 25 units. Each unit that is recalled by the participant either verbatim or as an acceptable paraphrase receives 1 point correct.
  The Delayed Recall score is the total points correct, and can range from 0 to 25. A higher value reflects a better outcome.
  units on a scale | 6.3 (2.1) | 8.8 (3.4) | 7.3 (2.6) | 7.4 (2.9)
Baseline Global Cognitive Function, as Measured by the Montreal Cognitive Assessment total score [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is a brief measure of global cognitive function. The total score has a range of 0 to 30; higher values represent a better outcome. Population: Two participants did not complete the measure due to lack of time (1, Active DLPFC) and pandemic disruption (1, Sham).
  units on a scale
    number analyzed (Participants) | 13 | 12 | 10 | 35
    (all) | 23.6 (4.6) | 23.9 (3.6) | 23.9 (2.7) | 23.8 (3.7)
Baseline Depressive Symptoms, as Measured by the Geriatric Depression Scale Total Score [Mean (Standard Deviation); unit: units on a scale] — The 15-item Geriatric Depression Scale (GDS) was used to screen for symptoms of depression. Five of the GDS items are oriented toward the absence of depressive symptoms (e.g., Do you feel full of energy?) and 10 are oriented toward current depressive symptoms (e.g., Do you often feel helpless?). The participant is asked to answer "yes" or "no" on the basis of how they have been feeling over the past week.
  The GDS total score ranges from 0 to 15. Lower values represent a better outcome.
  units on a scale | 2.6 (1.6) | 1.6 (1.3) | 2.9 (1.3) | 2.4 (1.5)
Total number of words correctly recalled, List Learning, California Verbal Learning Test-II [Mean (Standard Deviation); unit: total number of words correctly recalled] — The California Verbal Learning Test, Second edition (CVLT-II) is a memory task that yields several indices of the ability to learn a list of semantically related words and remember the list after a delay interval.
  The target list ("List A") of the CVLT-II contains 16 words. There are 5 orally presented learning trials; each is followed by immediate recall of the words in any order. The total number of words correctly recalled on the 5 list-learning trials was computed (range = 0 to 80). Higher values represent a better outcome.
  total number of words correctly recalled | 36.1 (10.5) | 47.0 (10.2) | 39.7 (11.2) | 40.7 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Words Correctly Recalled, List Learning, California Verbal Learning Test-II, Assessed 1 Week After Intervention and Adjusted for Baseline Performance
Description: The California Verbal Learning Test, Second edition (CVLT-II) is a memory task that yields several indices of the ability to learn a list of semantically related words and remember the list after a delay interval. The target list ("List A") of the CVLT-II contains 16 words.
  There are 5 orally presented learning trials; each is followed by immediate recall of the words in any order. The total number of words correctly recalled on the 5 list-learning trials was computed (range = 0 to 80). Higher values represent a better outcome.
Time Frame: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention.
Population: The population analyzed included all participants who received at least 1 session of the intervention and who provided primary outcome data at the 1-week primary endpoint.
Measure: Mean (Standard Deviation); unit: total number of words correctly recalled
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 14 | 12 | 11
total number of words correctly recalled | 36.1 (11.0) | 48.8 (8.7) | 37.0 (11.4)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); Test type: Superiority; p = 0.63, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-4.8 to 7.9], Standard Error of Mean 3.1
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); Test type: Superiority; p = 0.0476, Regression, Linear; Mean Difference (Final Values) = 6.9, 95% CI 2-sided [0.1 to 13.7], Standard Error of Mean 3.3

2. Secondary Outcome: Total Number of Words Correctly Recalled, List Learning, California Verbal Learning Test-II, Assessed 3 Months After Intervention and Adjusted for Baseline Performance
Description: as for outcome 1
Time Frame: 3 months after completing the 20-session intervention (acceptable window for assessment: 76-104 days after the final intervention session)
Population: The population analyzed included all participants who received at least 1 session of the intervention and who provided outcome data at the 3-month follow-up endpoint.
Measure: Mean (Standard Deviation); unit: total number of words correctly recalled
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 12 | 11 | 9
total number of words correctly recalled | 38.4 (10.3) | 53.0 (14.3) | 41.3 (6.9)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.45, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-11.4 to 5.2], Standard Error of Mean 4.1
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.21, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [-3.3 to 14.8], Standard Error of Mean 4.4

3. Secondary Outcome: California Verbal Learning Test-II (CVLT-II) Semantic Clustering Score, 1 Week After Intervention and Adjusted for Baseline Performance
Description: The California Verbal Learning Test, Second edition (CVLT-II) is a memory task that yields several indices of the ability to learn a list of 16 semantically related words and remember the list after a delay interval. There are 5 orally presented learning trials; each is followed by immediate recall of the words in any order.
  A measure of semantic clustering is calculated by a computer program. It is a measure of the participant's tendency to recall words in semantically organized clusters (e.g. the participant recalled "apple" and "orange" even though the two fruit words were not presented sequentially). The computer algorithm includes words recalled on Trials 1-5 and adjusts for the possibility that a semantic cluster occurred by chance. The range of CVLT-II Semantic Clustering Scores is -3 to 9. Higher values represent a better outcome.
Time Frame: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention.
Population: The population analyzed included all participants who received at least 1 session of the intervention and who provided outcome data at the 1-week endpoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 14 | 12 | 11
score on a scale | 0.5 (1.0) | 0.5 (1.2) | 0.1 (0.6)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.29, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-0.36 to 1.19], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.51, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.55 to 1.08], Standard Error of Mean 0.40

4. Secondary Outcome: Total Number of Words Correctly Recalled During the "Long Delay Free Recall" Component of the California Verbal Learning Test-II (CVLT-II), Assessed 1 Week After Intervention and Adjusted for Baseline Performance
Description: The California Verbal Learning Test, Second edition (CVLT-II) is a memory task that yields several indices of the ability to learn a list of semantically related words and remember the list after a delay interval. The target list ("List A") of the CVLT-II contains 16 words.
  After 5 learning trials and a subsequent 20-minute delay filled with unrelated tests, the participant was asked to recall the 16-word target list of the CVLT-II again. The total number of words correctly recalled was computed (range = 0 to 16). Higher values represent a better outcome.
Time Frame: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: total number of words correctly recalled
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 14 | 12 | 11
total number of words correctly recalled | 6.2 (4.2) | 10.3 (3.6) | 6.2 (3.5)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = .33, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-1.0 to 3.0], Standard Error of Mean 1.0
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.0038, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [1.1 to 5.3], Standard Error of Mean 1.0

5. Secondary Outcome: Depressive Symptoms, as Measured by the Geriatric Depression Scale (GDS), Assessed 1 Week After Intervention and Adjusted for Baseline Performance
Description: The 15-item Geriatric Depression Scale (GDS) was also used as an outcome measure. Five of the GDS items are oriented toward the absence of depressive symptoms (e.g., Do you feel full of energy?) and 10 are oriented toward current depressive symptoms (e.g., Do you often feel helpless?). The participant is asked to answer "yes" or "no" on the basis of how they have been feeling over the past week.
  The GDS total score ranges from 0 to 15. Lower values represent a better outcome.
Time Frame: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 14 | 12 | 11
score on a scale | 3.2 (2.3) | 1.9 (1.2) | 2.9 (2.3)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.58, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-1.1 to 2.0], Standard Error of Mean 0.78
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); Test type: Superiority; p = 0.59, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-2.2 to 1.3], Standard Error of Mean 0.86

6. Secondary Outcome: Everyday Functional Outcomes, as Measured by the Everyday Cognition (ECog) Questionnaire (Participant Version) Completed 1 Week After Intervention
Description: The Everyday Cognition (ECog) questionnaire is comprised of 39 items about the ability to perform everyday tasks. Each item relates to memory, language, visual-spatial, or executive function. Each item is rated on a scale from 1 to 4 (1 = better or no change…4 = consistently much worse compared to 10 years ago).
  For the Participant version of the ECog, the participant is asked to "Please rate your ability to perform certain everyday tasks now, as compared to your ability to do these same tasks 10 years ago." Total score range: 39-156. Higher values represent a worse outcome. The outcome score was adjusted for baseline.
Time Frame: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 11 | 12 | 11
score on a scale | 84.8 (21.0) | 66.1 (12.7) | 72.3 (16.1)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.30, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [-5.2 to 16.1], Standard Error of Mean 5.2
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.34, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-14.9 to 5.3], Standard Error of Mean 4.9

7. Secondary Outcome: Everyday Functional Outcomes, as Measured by the Everyday Cognition Questionnaire (Informant /Study Partner Version) Completed 1 Week After Intervention
Description: The Everyday Cognition (ECog) questionnaire is comprised of 39 items about the ability to perform everyday tasks. Each item relates to memory, language, visual-spatial, or executive function. Each item is rated on a scale from 1 to 4 (1 = better or no change…4 = consistently much worse compared to 10 years ago).
  For the Informant version of the ECog, the participant's study partner was asked to "Please rate the participant's ability to perform certain everyday tasks NOW, as compared to his/her ability to do these same tasks 10 years ago." Total score range: 39-156. Higher values represent a worse outcome. The outcome score was adjusted for baseline.
Time Frame: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention
Population: The population analyzed included the study partners of all participants who received at least 1 session of the intervention and whose study partner provided outcome data at the 1-week endpoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 12 | 9 | 5
score on a scale | 73.2 (30.9) | 61.1 (17.4) | 61.5 (29.2)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.996, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-22.0 to 22.1], Standard Error of Mean 10.6
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.87, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-20.6 to 24.3], Standard Error of Mean 10.8

8. Secondary Outcome: Instrumental Activities of Daily Living (IADLs), as Measured by the Functional Assessment Questionnaire, Completed 1 Week After Intervention
Description: Functional Assessment Questionnaire, completed by the study partner at end of treatment (1 week after intervention, adjusted for baseline). Each 10 item is rated on a scale from 0 to 3 (0 = Normal; 1 = Has difficulty, but does by self; 2 = Requires assistance; 3 = Dependent.
  Total score range: 0-30 (sum of 10 items). Interpretation: A total score of 9 (dependent in 3 or more activities) is the recommended cut-point for an indication of impaired function.
  Higher values represent a worse outcome.
Time Frame: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention.
Population: The population analyzed included the study partners of all participants who received at least 1 session of the intervention and whose study partners provided outcome data at the 1-week endpoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 14 | 9 | 6
score on a scale | 3.29 (4.41) | 1.00 (1.32) | 1.33 (3.27)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.97, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-2.14 to 2.22], Standard Error of Mean 1.06
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.91, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-2.15 to 2.41], Standard Error of Mean 1.11

9. Secondary Outcome: Global Cognitive Function, as Measured by the Montreal Cognitive Assessment (MoCA), Assessed 1 Week After Intervention and Adjusted for Baseline
Description: The Montreal Cognitive Assessment (MoCA) is a brief measure of global cognitive function. The total score has a range of 0 to 30; higher values represent a better outcome.
Time Frame: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 11 | 11 | 10
score on a scale | 23.0 (4.5) | 23.8 (2.8) | 23.6 (2.2)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.84, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-2.3 to 1.9], Standard Deviation 1.0
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.80, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-1.9 to 2.4], Standard Error of Mean 1.0

10. Secondary Outcome: Visuospatial Memory, as Measured by the Brief Visuospatial Memory Test-Revised (BVMT-R), assessed1 Week After Intervention and Adjusted for Baseline Performance
Description: Brief Visuospatial Memory Test-Revised (BVMT-R) Trials 1-3 total recall raw score at end of treatment (1 week after intervention, adjusted for baseline); range: 0-36; higher values represent a better outcome
Time Frame: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 12 | 11 | 10
score on a scale | 17.8 (8.5) | 18.5 (6.2) | 21.6 (6.5)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.48, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-5.5 to 2.6], Standard Error of Mean 2.0
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.18, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-6.8 to 1.3], Standard Error of Mean 2.0

11. Secondary Outcome: Language Function, as Measured by Category Fluency (CF), Assessed 1 Week After Intervention and Adjusted for Baseline Performance
Description: Category Fluency is a measure of verbal fluency in which the participant is asked to generate different exemplars from a semantic category specified by the examiner. For example, if the examiner says, 'articles of clothing,' correct responses include exemplars such as, 'shirt,' 'tie,' or 'hat.' The participant is given one minute to say all the responses they can think of. The values reported reflect the total number of correct, unique responses produced. Higher values represent a better outcome.
Time Frame: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: correct, unique responses
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 14 | 12 | 11
correct, unique responses | 16.7 (3.8) | 19.8 (4.8) | 19.4 (6.0)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.075, Regression, Linear; Adjusted for baseline; Median Difference (Final Values) = -2.7, 95% CI 2-sided [-5.7 to 0.3], Standard Error of Mean 1.5
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.195, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-5.4 to 1.1], Standard Error of Mean 1.6

12. Secondary Outcome: Language Function, as Measured by 42-item Boston Naming Test (BNT), Assessed 1 Week After Intervention and Adjusted for Baseline Performance
Description: The Boston Naming Test (BNT) assesses the ability to verbally name pictured objects. The subject is shown a series of line drawings and asked to name the object. The test items become progressively more difficult. (The 42 items are presented in order of decreasing frequency of the target word). The total number of correct responses can range from 0 to 42. Higher values represent a better outcome.
Time Frame: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 11 | 11 | 10
correct responses | 36.3 (3.9) | 38.4 (3.8) | 35.9 (4.8)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.28, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-1.0 to 3.4], Standard Error of Mean 1.1
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.21, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-0.8 to 3.6], Standard Error of Mean 1.1

13. Secondary Outcome: Visuoconstructional Function, as Measured by the Rey-Osterrieth Complex Figure (ROCF) Copy Score, assessed1 Week After Intervention and Adjusted for Baseline Performance.
Description: Rey-Osterrieth Complex Figure (ROCF) Copy score at end of treatment (1 week after intervention, adjusted for baseline); range: 0-36; higher values represent a better outcome
Time Frame: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 12 | 11 | 10
score on a scale | 33.8 (4.1) | 32.7 (3.8) | 34.9 (1.8)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.66, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-3.2 to 2.1], Standard Error of Mean 1.3
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.11, Regression, Linear; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-4.9 to 0.5], Standard Error of Mean 1.3

14. Secondary Outcome: Speed of Processing and Executive Function, as Measured by Trail Making Part B, Assessed 1 Week After Intervention and Adjusted for Baseline Performance
Description: In the Trail Making Part B test, the response form has a series of 25 circles; each circle contains a number or a letter. The participant is asked to connect the circles in order by alternating between the numbers and letters. The maximum time allowed is 300 seconds. Trails B is thought to require executive skills as well as processing speed. The Trail Making B seconds-to-complete scores were log transformed because the distribution of scores was positively skewed. We also reverse scored the log scores so that higher values would indicate a better outcome. To reverse the log scores, we used the formula:
  reverse score = max(x) + 1 - x, where max(x) is the natural log of 300 or 5.70378.
  For example, if a participant's time-to-complete score was 74 seconds, the natural log transformed score was 4.304. Reverse scoring yields a value of 2.4 (2.4 = 5.70378 + 1 - 4.304). The reverse-scaled, log transformed seconds-to-complete scores were used in all statistical analyses.
Time Frame: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: reverse scaled, log transformed scores
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 12 | 11 | 10
reverse scaled, log transformed scores | 2.11 (0.64) | 2.42 (0.32) | 2.42 (0.33)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.59, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.29 to 0.17], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); a priori threshold for statistical significance = .05; Test type: Superiority; p = 0.64, Regression, Linear; Adjusted for baseline; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.17 to 0.28], Standard Error of Mean 0.11

15. Secondary Outcome: Attention, as Measured by the Attentional Network Task (ANT), Assessed 1 Week After Intervention and Adjusted for Baseline Performance
Description: Attentional Network Task(ANT) correct reaction time, as measured by the ANT computerized test
Time Frame: planned: 1 week after completing the 20-session intervention, which was typically 4 weeks after starting the intervention.
Population: There are no data to report in the Outcome Measure Data Table because the protocol was modified (i.e., amended) to not administer the Attention Network Task. The amendment can be found on page 63 of the updated Study Protocol and Statistical Analysis Plan, dated 09/19/2019.
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Change From Baseline in Brain Functional Connectivity
Description: Change from Baseline in Functional connectivity metrics (derived from the pre- and the post-intervention functional magnetic resonance imaging (fMRI) scans rs-fMRI scans) will be computed with respect to: connectivity within the Default Mode Network (DMN), and connectivity between the DMN and the Central Executive Network (CEN).
Time Frame: as for outcome 15
Population: Data cannot be reported because change from Baseline in Functional connectivity metrics required post-intervention resting-state functional magnetic resonance imaging (fMRI) scan data that could not be acquired after March of 2020 due to COVID-19 suspension of in-person research and subsequent early termination of the NIA award in August of 2021.
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Pre-post Change in Peripheral Levels of Brain-derived Neurotrophic Factor (BDNF)
Description: Brain-derived Neurotrophic Factor (BDNF) plasma levels were measured from blood samples that were collected during the first session and the last session of TMS intervention, after a minimum of 4 hours of fasting.
  Higher change scores represent a better outcome.
Time Frame: First Intervention session to Last Intervention session. The average time frame from the first to the 20th and last session is 18 days.
Population: All participants who had BDNF plasma results for both pre- and post-intervention, i.e. during the first session and the last session of TMS.
  Additional comments: (1) All of these participants were treatment adherent per study protocol, i.e., they completed at least 18 of the 20 rTMS sessions. (2) All of these participants provided behavioral outcome data at the primary endpoint, i.e. 1 week after completion of the TMS intervention.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
Number analyzed (Participants) | 12 | 10 | 9
pg/mL | 394.83 (1773.65) | 1188.85 (3513.12) | 687.17 (2145.18)
Statistical Analysis 1: Comparison: Active rTMS (Bilateral DLPFC) vs Active rTMS (Bilateral LPC) vs Placebo rTMS (Inactive); Test type: Superiority; p = 0.768, ANOVA — a priori threshold for statistical significance = .05

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from over a period of 6 to 12 months. The reporting timeframe for All-Cause Mortality and Serious Adverse Events is from enrollment and randomization until 6 months after completion of the 20-session device intervention, typically 7 months. The reporting timeframe for other adverse events is from enrollment and randomization until 1 week after completion of the 20-session device intervention, typically 1 month.
Description: Medical Dictionary for Regulatory Activities (MedDRA)
Arm/Group | Active rTMS (Bilateral DLPFC) | Active rTMS (Bilateral LPC) | Placebo rTMS (Inactive)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/13 | 2/13
Other Adverse Events (participants affected / at risk) | 5/14 | 5/13 | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (Bilateral DLPFC) (N=14) | Active rTMS (Bilateral LPC) (N=13) | Placebo rTMS (Inactive) (N=13)
pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
rotator cuff (surgerical repair) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (Bilateral DLPFC) (N=14) | Active rTMS (Bilateral LPC) (N=13) | Placebo rTMS (Inactive) (N=13)
Site discomfort (General disorders) | 3 (3) | 2 (2) | 0 (0) — Organ System full name: General disorders and administration site conditions
Toothache/TMJ pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Muscle twitching of left jaw
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) — Organ System full name: General disorders and administration site conditions
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Smaller numbers of subjects were enrolled than originally proposed. Reasons included: a protracted start-up, low enrollment during Years 1 and 2, the cessation of TMS intervention visits and new enrollment during the COVID-19 pandemic in Year 3, and National Institute on Aging's decision to terminate the award in Year 4.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT03331796/Prot_SAP_002.pdf